CLINICAL TRIAL: NCT02497170
Title: Implementation of A Patient Centered Self-Management Program for Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO201500001877
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Life style changes (Other): Pre and post after education intervention Education program
  Interventions: Behavioral: Education of goal setting and achievement

INTERVENTIONS:
Behavioral: Education of goal setting and achievement — Education of American Association of Diabetes Educations 7 behavioral goals and how to achieve them

SUMMARY:
Translational study based on the American Association of Diabetes Educators 7 behaviors to manage Type 2 diabetes

DETAILED DESCRIPTION:
The Primary Investigator will meet with patients that attend routine visits for Diabetes 2 in the primary care office on a monthly basis to set behavior goals. Behavior goals will be set by patient's choice of 4 out of 7 of the AADE7 recommendations. The goals are health eating, being active, monitoring,taking medications, problem solving, healthy coping, and reducing risk. Once the goal is chosen, the PI and patient will make a plan to address the goals on a monthly basis for four months. There will be pre and post questionnaires that will evaluate diabetes knowledge and self-efficacy. There will also be a pre and post measure of the patient's Hemoglobin A1c which is a measurement that helps determine the extent of glycemic control over a three-month period.

The goal of the study is to determine if translation of the AADE7 behavioral goals into the primary care setting will make a difference in diabetes knowledge, self efficacy, and Hemoglobin A1c.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 with Hemoglobin A1c 7 mmol/mol or higher will be included in the study
* Patients willing to attend minimum of 4 monthly appointments for diabetes treatment
* Patients who give written consent to participate

Exclusion Criteria:

* Patients below age 18, children are not treated in the facility for type 2 diabetes
* Patients who attend less than 4 monthly appointments for diabetes,
* Patients who do no give written consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 4 months
  Pre and Post Differences

CONTACTS AND LOCATIONS:
Overall Officials: melissa souza, Principal Investigator — Rutgers University Newark New Jersey
Locations (1):
- Melissa Souza, Somerdale, New Jersey, United States